CLINICAL TRIAL: NCT03579524
Title: The Effectiveness of Pain Relieve of Ultrasound-guided Erector Spinae Plane Block Versus Serratus Anterior Plane Block With General Anesthesia in Modified Radical Mastectomy Patient (Randomized Double-Blinded Controlled Clinical Trial)
Brief Title: Comparison of Erector Spinae Plane Block With Serratus Anterior Plane Block for Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Hany M Yassin, MD, Associated professor, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: M336
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Pain; Breast Cancer
Keywords: Erector Spinae Plane Block; Serratus Anterior Plane Block
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Active Comparator): Erector Spinae Plane Block administered group
  Interventions: Procedure: Erector Spinae Plane Block
- SAPB group (Active Comparator): Serratus Anterior Plane Block administered group
  Interventions: Procedure: Serratus Anterior Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — At lateral decubitus with the operation site up, the vertebrae will be counted from cephalad to caudal direction until reaching T5 spinous process as the first palpable spinous process is C7. The ultrasound probe will be placed vertically 3 cm lateral to the T5 spinous process. Three muscles will be identified superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. The needle will be introduced from superior to inferior direction in-plane until the tip lay deep to erector spinae muscle. 0.5: 1 mL of non-active fluid will be injected to confirm correct needle tip position by visualizing spread under erector spinae muscle. A total of 20 mL of 0.25% bupivacaine will be injected next.
  Other Names: ESPB
  Arms: ESPB group
Procedure: Serratus Anterior Plane Block — At supine position with the arm abducted, the ribs will be counted in the mid-axillary line from downward upwards until the 5th ribs. The linear probe will be placed horizontally then three muscles will be identified: latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscles (deep and inferior). The needle will be inserted in-plane with respect to the ultrasound probe from supero-anterior to posteroinferior. 0.5: 1 mL of non-active fluid will be injected to confirm correct needle tip position by visualizing spread over serratus anterior muscles, then a total 20 ml of bupivacaine 0.25% will be injected.
  Other Names: SAPB
  Arms: SAPB group

SUMMARY:
Breast cancer is by far the world's most common cancer among women and the most common cause of female death from cancer worldwide. It's worldwide incidence is 43.4 in 100.000 while in Egypt is 48.8 in 100.000.

One of the most common surgical procedures for it is modified radical mastectomy (MRM), It is account for 31% of all breast surgery cases.

Post-mastectomy pain is a big problem affecting the outcome of surgery. It was used to be managed by opioids which may lead to many side effects such as nausea, vomiting, ileus, over sedation and respiratory depression. Chronic pain syndrome (phantom breast pain, paraesthesias, and intercostobrachial neuralgia) may be developed due to inadequate pain control.

So many regional analgesic techniques have been developed for effective pain control.

The safest and easiest is local wound infiltration with local anesthesia but the duration of action is limited. Intercostal nerve block and interpleural block are effective, but there is a fear of pneumothorax and transient Horner's syndrome.

Thoracic epidural analgesia is not preferred however it's efficacy because of possible neurological and hemodynamic side effects.

The gold standard now is thoracic paravertebral block (PVB) which provide effective analgesia with minimal hemodynamic derangement but it carries a risk of pneumothorax in addition to slightly complex technique.

Ultrasound-guided interfascial plane blocks such as pectoral nerve (PECS) block type 1 and 2 , serratus anterior plane block (SAPB) and erector spinae plane block (ESP) which is a recent block newly described for various surgeries for postoperative analgesia have also been reported as alternatives, with the advantages of simplicity, ease of performance and fewer complications.

there is no sufficient Randomized controlled trails that assess the effectiveness and safety of erector spinae plane block ESPB in controlling post mastectomy pain This study compares the analgesic efficacy of ultrasound-guided erector spinae plane block (ESPB) and serratus anterior plane block (SAPB) in patients undergoing MRM with axillary dissection.

DETAILED DESCRIPTION:
Preoperative preparation:

History taking, physical examination, and investigations will be done according to the local protocol designed to evaluate the patients. This includes complete blood count, blood sugar level, serum urea and creatinine, liver function tests, coagulation profile and electrocardiogram (ECG).

Before surgery, the participants will receive education about the VAS pain score (0-100 mm) (where0=no pain and 100 = worst comprehensible pain) and the details of the nerve block procedures. After 6 hours of fasting, the patients will be taken to the operation theatre.

Anesthetic management:

The patient will receive Midazolam 0.03 mg/kg intravenous (IV), Metoclopramide 10 mg IV, Ranitidine 50 mg IV and Cefotaxime 1 gm as a premedication.

Intravenous access will be obtained with an 18-gauge intravenous (IV) cannula in the contralateral upper limb of the surgical site and monitors (pulse oximeter, electrocardiography, non-invasive blood pressure (NIBP) and capnography) will be applied.

All patients will receive pre-oxygenation with 100% O2 for 3 min. Anesthesia will be induced by using fentanyl 1μg/kg, propofol 1.5-2 mg/kg and atracurium 0.5 mg/kg. Anesthesia will be maintained by controlled ventilation with oxygen and air (50:50) with target of End Tidal Carbon Dioxide Tension (EtCO2) ≈ 35-40 mmHg, isoflurane 1:1.5 minimum alveolar concentration (MAC), 0.5μg/kg fentanyl will be given intraoperatively when either heart rate or Non-Invasive Blood Pressure (NIBP) report an increase by more than 20% of the basal records. Anesthesia will be discontinued and tracheal extubation will be done once patient fulfilled the extubation criteria.

A high-frequency ultrasound probe Active Array L12-4 (8-13MHz) of an ultrasound machine (Philips clear vue350, Philips Healthcare, Andover MA01810™, USA).and a 22-gauge, 50 mm echogenic needle (Stimuplex D®; B Braun, Germany) will be used for performing the blocks.

Patients in group (S) will receive serratus anterior plane block and those in group (E) will receive Erector spinae plane block. Both of these blocks will be performed after induction of general anesthesia by an experienced anesthesiologist (who is well trained in ultrasound-guided regional anesthesia). After proper skin sterilization with povidone-iodine solution.

For the ultrasound-guided serratus anterior plane block, the patient will be placed in supine position with the arm abducted. Ribs will be counted in the mid-axillary line from downward upwards until the 5th ribs the linear probe will be placed horizontally then three muscles will be identified: latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscles (deep and inferior) .the thoracodorsal artery (slightly posterior) will be used as extra guide in the identification of the plane superficial to the serratus muscle. The needle will be inserted in-plane with respect to the ultrasound probe from supero-anterior to postero-inferior. 0.5: 1 mL of non-active fluid will be injected to confirm correct needle tip position by visualizing spread over serratus anterior muscles, then a total 20 ml of bupivacaine 0.25% will be injected.

For the ultrasound-guided erector spinae plane block

At first the patient will be placed in a lateral decubitus with the operation site up. The vertebrae will be counted from cephalad to caudal direction until we reach T5 spinous process as the first palpable spinous process is C7. Ultrasound probe will be placed vertically 3 cm lateral to the T5 spinous process. Three muscles will be identified superficial to the hyperechoic transverse process shadow as follows:

trapezius, rhomboid major, and erector spinae. The needle will be introduced from superior to inferior direction in-plane until the tip lay deep to erector spinae muscle (the needle tip contacts the tip of the transverse process), 0.5: 1 mL of non-active fluid will be injected to confirm correct needle tip position by visualizing spread under erector spinae muscle a total of 20 mL of 0.25% bupivacaine will be injected next.

Post-operative care Patients will be transferred to post-anesthetic care unit (PACU) for 2 hrs after anesthesia emergence. The patients will be discharged from the PACU after fulfilling the discharge criteria based on the modified Aldrete score> 9 The patient will receive analgesic according to the local institutional protocol as the following (paracetamol 1gm IV infusion/8 hours, ketorolac 30 mg Intramuscular/12 hours) as 2 components of multimodal anesthesia regimen for postoperative pain control.

A postoperative rescue analgesia with morphine sulfate IV per a titration protocol (3 mg IV as a bolus dose which can be repeated every 5 minutes with a maximum dose of 15mg per 4 hours or 45mg per 24 hours) will be employed if visual analog pain scale (VAS) > 4. The morphine titration protocol will be suspended with Oxygen saturation < 95%; Respiratory rate < 10 / min; the development of sedation (Ramsay sedation scale >2); development of acute adverse effects (allergy, marked itching, excessive vomiting, and hypotension with systolic blood pressure less than 20% of baseline values); or attaining adequate level of analgesia.

ELIGIBILITY:
Inclusion Criteria:

* female aged >18 years with breast cancer eligible for modified radical mastectomy.
* American Society of Anesthesiologists Physical Status I to IV.

Exclusion Criteria:

* Patient refusal.
* body mass index (BMI) > 40.
* local infection at the site of the block.
* local anesthetic allergy.
* significant neurological or respiratory disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Patient with Breast Cancer
Enrollment: 62 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
The duration of analgesia of the two blocks | At 48 hours postoperative
  the pain will be assisted based on the time needed for the first dose rescue analgesia.

SECONDARY OUTCOMES:
The cumulative opioids (morphine) consumption | At 24 hours postoperative
  The total amount of opioids received post operative
The cumulative opioids (morphine) consumption | At 48 hours postoperative
  The total amount of opioids received post operative
The intervals between opioid (morphine) doses | At 24 hours postoperative
  the time needed between two successive opioid doses
The intervals between opioid (morphine) doses | At 48 hours postoperative
  the time needed between two successive opioid doses
The quality of analgesia based on visual analogue scale (VAS) pain score at rest | At one hour postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at rest | At 6 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at rest | At 12 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at rest | At 18 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at rest | At 24 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at rest | At 30 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at rest | At 36 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at rest | At 42 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at rest | At 48 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at arm abduction | At one hour postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at arm abduction | At 6 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at arm abduction | At 12 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at arm abduction | At 18 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at arm abduction | At 24 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at arm abduction | At 30 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at arm abduction | At 36 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at arm abduction | At 42 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
The quality of analgesia based on visual analogue scale (VAS) pain score at arm abduction | At 48 hours postoperative
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
Incidences of complications related to both techniques | up to 72 hours postoperative
  complications related to the Block or drug administered
Nausea | At 2 hours postoperative
  Morphine related side effect
Nausea | At 6 hours postoperative
  Morphine related side effect
Nausea | At 12 hours postoperative
  Morphine related side effect
Nausea | At 24 hours postoperative
  Morphine related side effect
Nausea | At 48 hours postoperative
  Morphine related side effect
Nausea | At 72 hours postoperative
  Morphine related side effect
Vomiting | At 2 hours postoperative
  Morphine related side effect
Vomiting | At 6 hours postoperative
  Morphine related side effect
Vomiting | At 12 hours postoperative
  Morphine related side effect
Vomiting | At 24 hours postoperative
  Morphine related side effect
Vomiting | At 48 hours postoperative
  Morphine related side effect
Vomiting | At 72 hours postoperative
  Morphine related side effect
Pruritus | At 2 hours postoperative
  Morphine related side effect
Pruritus | At 6 hours postoperative
  Morphine related side effect
Pruritus | At 12 hours postoperative
  Morphine related side effect
Pruritus | At 24 hours postoperative
  Morphine related side effect
Pruritus | At 48 hours postoperative
  Morphine related side effect
Pruritus | At 72 hours postoperative
  Morphine related side effect
Over-sedation | At 2 hours postoperative
  Morphine related side effect
Over-sedation | At 6 hours postoperative
  Morphine related side effect
Over-sedation | At 12 hours postoperative
  Morphine related side effect
Over-sedation | At 24 hours postoperative
  Morphine related side effect
Over-sedation | At 48 hours postoperative
  Morphine related side effect
Over-sedation | At 72 hours postoperative
  Morphine related side effect
Urine retension | At 2 hours postoperative
  Morphine related side effect
Urine retension | At 6 hours postoperative
  Morphine related side effect
Urine retension | At 12 hours postoperative
  Morphine related side effect
Urine retension | At 24 hours postoperative
  Morphine related side effect
Urine retension | At 48 hours postoperative
  Morphine related side effect
Urine retension | At 72 hours postoperative
  Morphine related side effect
The duration of surgery | Once at completion of surgery
  time needed to perform surgery
Intraoperative fentanyl needed | Once at completion of surgery
  The amount of Fentanyl given intraoperative as fentanyl will be given when either heart rate or NIBP(Non-Invasive Blood Pressure) report an increase by more than 20% of the basal records
Patients' satisfaction with postoperative analgesia | after 72 hours postoperative
  Will be evaluated according to a satisfaction score (poor = 0; fair = 1; good = 2; excellent= 3)
Age | Once the patient is recruited
  In years
weight | Once the patient is recruited
  In kilograms
Height | Once the patient is recruited
  In meters
BMI | Once the patient is recruited
  In kilogram per square meter

CONTACTS AND LOCATIONS:
Overall Officials: Hany M. Yassin, MD, Principal Investigator — Fayoum University Hospitals; Mohamed A. Shawky, MD, Study Chair — Fayoum University Hospital
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonvicini D, Giacomazzi A, Pizzirani E. Use of the ultrasound-guided erector spinae plane block in breast surgery. Minerva Anestesiol. 2017 Oct;83(10):1111-1112. doi: 10.23736/S0375-9393.17.12015-8. Epub 2017 May 11. No abstract available. PMID 28492298
- [Background] Bonvicini D, Tagliapietra L, Giacomazzi A, Pizzirani E. Bilateral ultrasound-guided erector spinae plane blocks in breast cancer and reconstruction surgery. J Clin Anesth. 2018 Feb;44:3-4. doi: 10.1016/j.jclinane.2017.10.006. Epub 2017 Oct 21. No abstract available. PMID 29065335
- [Background] Veiga M, Costa D, Brazao I. Erector spinae plane block for radical mastectomy: A new indication? Rev Esp Anestesiol Reanim (Engl Ed). 2018 Feb;65(2):112-115. doi: 10.1016/j.redar.2017.08.004. Epub 2017 Nov 2. English, Spanish. PMID 29102405
- [Background] Kimachi PP, Martins EG, Peng P, Forero M. The Erector Spinae Plane Block Provides Complete Surgical Anesthesia in Breast Surgery: A Case Report. A A Pract. 2018 Oct 1;11(7):186-188. doi: 10.1213/XAA.0000000000000777. PMID 29688930
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Matsumoto M, Flores EM, Kimachi PP, Gouveia FV, Kuroki MA, Barros ACSD, Sampaio MMC, Andrade FEM, Valverde J, Abrantes EF, Simoes CM, Pagano RL, Martinez RCR. Benefits in radical mastectomy protocol: a randomized trial evaluating the use of regional anesthesia. Sci Rep. 2018 May 18;8(1):7815. doi: 10.1038/s41598-018-26273-z. PMID 29777144
- [Background] Gupta K, Srikanth K, Girdhar KK, Chan V. Analgesic efficacy of ultrasound-guided paravertebral block versus serratus plane block for modified radical mastectomy: A randomised, controlled trial. Indian J Anaesth. 2017 May;61(5):381-386. doi: 10.4103/ija.IJA_62_17. PMID 28584346